CLINICAL TRIAL: NCT01502631
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of SUN13837 Injection in Adult Subjects With Acute Spinal Cord Injury
Brief Title: Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of SUN13837 Injection in Adult Subjects With Acute Spinal Cord Injury (ASCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASBI 603
Record Dates: First submitted 2011-12-27; First posted 2012-01-02 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Acute Spinal Cord Injury
Keywords: ASCI; SUN13837; Acute traumatic cervical spinal cord injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SUN13837 (Active Comparator)
  Interventions: Drug: SUN13837 injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUN13837 injection — SUN13837 injection, injection 1 x daily for 28 doses
  Arms: SUN13837
Drug: Placebo — Matching placebo, volume equivalent to injection 1 x daily for 28 doses
  Arms: Placebo

SUMMARY:
The purpose of this research study is to gather scientific information about the effectiveness of the study drug, SUN13837 Injection, when compared with the placebo (inactive substance) in participants with acute spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Acute traumatic injury to the cervical neurological spinal cord as follows:

   1. American Spinal Injury Association Impairment Scale A (AIS A) with a level of injury at either cervical level C4, C5, C6, C7 (for C4, the participant must have at least 1 point of motor activity within the zone of partial preservation (ZPP) inclusive of C5 to thoracic level 1 [T1]). In addition, the AIS A participant may be included if ALL of the following are present 1) the most caudal intact sensory segment (both pinprick and light touch) is C3, 2) at least one side (right or left) has both intact pinprick and light touch sensation in the C4 dermatome, AND 3) at least 1 point of motor activity within the ZPP inclusive of C5 to T1
   2. American Spinal Injury Association Impairment Scale B or C (AIS B or C) with a neurological level of injury at either C3, C4, C5, C6, C7, or C8 AND a total LEMS of 5 or fewer motor points
2. Closed single traumatic spinal cord injury occurring within 12 hours of first dosing
3. Male or female cervical AIS A participants ≥ 16 to ≤ 80 years and male or female cervical AIS B or C participants ≥16 to ≤70 years
4. Females of childbearing potential and males must agree to maintain adequate contraception for the first 35 days of the study

Exclusion Criteria:

1. Unable to obtain informed consent (either from the participant or from the participant's legally authorized representative [LAR])
2. Women who are breastfeeding (if unwilling to stop for the first 35 days of the study) or who are pregnant
3. Coma or significant impairment in the level of consciousness that interferes with the performance or interpretation of protocol specified assessments
4. Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol specified assessments
5. Unable, as determined by the investigator, or unwilling to discontinue use of potent P-glycoprotein (P-gp) inhibitors for the first 35 days of the study
6. Unable, as determined by the investigator, or unwilling to discontinue use of potent cytochrome P450 (CYP) 3A4/5 inducers for the first 35 days of the study
7. Renal compromise (serum creatinine greater than 1.5 times the age- and sex-appropriate upper limit of normal [ULN]) at screening before the first dose of study drug
8. Severe Hepatic dysfunction (serum alanine transaminase [ALT], aspartate transaminase [AST], and/or gamma-glutamyltransferase [GGT] ALL greater than 2.5 times the age- and sex-appropriate ULN) or hepatic impairment (detectable ascites, serum bilirubin greater than 2 mg/dL, serum albumin less than 3.5 g/dL, and prothrombin time prolonged by more than 6 seconds above the ULN for the local laboratory in the absence of anticoagulant therapy) at screening before the first dose of study drug
9. Concomitant spinal cord injury or abnormality as determined by routine imaging:

   1. Conclusive radiological evidence of complete spinal cord transection
   2. Multiple injuries to the neurological spinal cord at different levels
10. History of symptomatic cervical spinal stenosis with myelopathy as a factor confounding participant assessment
11. Unlikely to be available for follow-up as specified in the protocol
12. Participated in a previous clinical study and received an investigational product within 30 days of screening
13. Previous exposure to SUN13837
14. Allergy to SUN13837 or any of its excipients
15. Any other issue which, in the opinion of the investigator, made the participant unsuitable for study participation.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2014-09-21 (Actual); Study Completion 2014-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (56):
- United States (35):
  - Tucson, Arizona
  - Downey, California
  - Los Angeles, California
  - Sacramento, California
  - San Jose, California
  - Denver, Colorado
  - Englewood, Colorado
  - Newark, Delaware
  - Hollywood, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Davenport, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Columbia, Missouri
  - Kansas City, Missouri
  - Springfield, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Camden, New Jersey
  - Newark, New Jersey
  - West Orange, New Jersey
  - Great Neck, New York
  - Stony Brook, New York
  - Valhalla, New York
  - White Plains, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Dayton, Ohio
  - Malvern, Pennsylvania
  - Philadelphia, Pennsylvania
  - Milwaukee, Wisconsin
- Canada (4):
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- Czechia (4):
  - Brno
  - Liberec
  - Ostrava
  - Prague
- France (5):
  - Amiens
  - Berck
  - Bordeaux
  - Lille
  - Montpellier
- Poland (2):
  - Lodz
  - Sosnowiec
- Spain (3):
  - A Coruña
  - Barcelona
  - Seville
- United Kingdom (3):
  - Edgbaston, Birmingham
  - Glasgow, Scotland
  - Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 19 clinic sites in the United States of America, 2 in France, 1 in the United Kingdom,1 in Spain, and 1 in the Czech Republic. Four (4) of the participants were not treated. The data on the 61 treated participants are presented in this report.
Pre-assignment Details: Participants with acute traumatic cervical spinal cord injury (ASCI) within 12 hours of treatment were enrolled in this study.
Groups:
- SUN13837: Participants with acute traumatic cervical spinal cord injury who were administered SUN13837 injection once daily for at least 7 but no more than 28 consecutive days (except for the dose interval between the first and second doses, which may have occurred on the same day [dosing to 27 days] in certain participants).
- Placebo: Participants with acute traumatic cervical spinal cord injury who were administered a placebo once daily for at least 7 but no more than 28 consecutive days (except for the dose interval between the first and second doses, which may have occurred on the same day [dosing to 27 days] in certain participants).
Period: Overall Study
Arm/Group | SUN13837 | Placebo
Started | 30 | 31
Completed | 10 | 11
Not Completed | 20 | 20
Not completed — Adverse Event | 5 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — Participant withdrew consent | 2 | 4
Not completed — Participant non-compliant | 1 | 0
Not completed — Investigator's decision | 0 | 1
Not completed — Other | 10 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | SUN13837 | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (16.6) | 38.8 (17.2) | 38.4 (16.8)
Age, Customized [Count of Participants; unit: Participants]
  < 55 years | 25 | 25 | 50
  ≥ 55 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 4 | 5 | 9
  White | 22 | 17 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Spinal Cord Independence Measure, Version III (SCIM III) Score Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord Injury
Description: The SCIM III is a comprehensive rating scale that measures the ability of participants with spinal cord injury to perform everyday tasks. The SCIM III has 19 items that assess 3 domains: Self-Care (6 items, scores range from 0 to 20), Respiration and Sphincter Management (4 items, scores range from 0 to 40), and Mobility (9 items, scores range from 0 to 40). The total SCIM score ranges from 0 to a maximum of 100 points in an individual with a fully functional spinal cord. A score of 0 indicates a worse outcome and a score of 100 indicates a better outcome. An improvement of at least 4 points of the total SCIM showed a small significant improvement, and 10 points showed a substantial improvement.
Time Frame: Week 2, week 4, week 8 and week 16 post dose.
Population: Total Spinal Cord Independence Measure was assessed in the intent-to-treat (ITT) population, defined as all randomized participants who had at least 1 SCIM III evaluation and received at least 7 (partial or complete) IV bolus dose injections of the study drug in SUN13837 group or in Placebo group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Score on a scale
  Week 2 | 15.87 [10.15 to 21.59] | 10.26 [4.73 to 15.79]
  Week 4 | 22.56 [15.65 to 29.47] | 15.69 [8.87 to 22.51]
  Week 8 | 28.77 [21.34 to 36.20] | 25.74 [18.39 to 33.09]
  Week 16 | 38.14 [30.14 to 46.14] | 33.60 [25.67 to 41.53]
Statistical Analysis 1: Comparison: SUN13837 vs Placebo; Difference (SUN13837 - Placebo) at Week 2; Test type: Superiority; p = 0.2182, Mixed Model Repeated Measures (MMRM); Least Squares (LS) Mean = 5.61, 90% CI 2-sided [-1.93 to 13.14], Standard Error of Mean 4.497
Statistical Analysis 2: Comparison: SUN13837 vs Placebo; Difference (SUN13837 - Placebo) at Week 4; Test type: Superiority; p = 0.2260, Mixed Model Repeated Measures (MMRM); Least Squares (LS) Mean = 6.87, 90% CI 2-sided [-2.54 to 16.27], Standard Error of Mean 5.583
Statistical Analysis 3: Comparison: SUN13837 vs Placebo; Difference (SUN13837 - Placebo) at Week 8; Test type: Superiority; p = 0.6184, Mixed Model Repeated Measures (MMRM); Least Squares (LS) Mean = 3.03, 90% CI 2-sided [-7.15 to 13.21], Standard Error of Mean 6.023
Statistical Analysis 4: Comparison: SUN13837 vs Placebo; Difference (SUN13837 - Placebo) at Week 16; Test type: Superiority; p = 0.4912, Mixed Model Repeated Measures (MMRM); Least Squares (LS) Mean = 4.54, 90% CI 2-sided [-6.48 to 15.56], Standard Error of Mean 6.524

2. Secondary Outcome: Sensitivity Analyses of Total Spinal Cord Independence Measure, Version III (SCIM III) Score at Week 16 by Treatment Group
Description: as for outcome 1
Time Frame: Week 16 post dose
Population: Sensitivity analyses were assessed in the Intent-to-Treat (ITT) and Efficacy Evaluable (EE) populations. The EE Population consisted of all subjects in the ITT Population who did not have any major protocol violations that impacted efficacy and were observed for efficacy for at least 2 SCIM III evaluations.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Score on a scale
  Primary (EE): number analyzed (Participants) | 24 | 25
  Primary (EE) | 38.25 [30.96 to 45.54] | 30.48 [23.41 to 37.55]
  LOCF (ITT) | 36.12 [28.60 to 43.64] | 30.84 [23.38 to 38.30]
  Multiple Imputation (ITT) | 37.96 [29.32 to 46.61] | 32.17 [23.46 to 40.88]
  Simple Multiple Imputation (ITT) | 38.49 [30.06 to 46.93] | 32.00 [23.63 to 40.38]

3. Secondary Outcome: Change From Baseline of Total Motor Score (TMS) of International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord Injury
Description: TMS was the sum of the overall Upper Extremity Motor Score (UEMS) and the overall Lower Extremity Motor Score (LEMS) of ISNCSCI. The score on the scale runs from a minimum value of 0 to a maximum of 100 points in an individual with a fully functional spinal cord. A score of 0 indicates a worse outcome and a score of 100 indicates a better outcome. The UEMS was defined as the sum of the motor function scores in the cervical spinal segments C5, C6, C7, C8, and T1. A separate sum was obtained for the right and left sides (a maximum of 25 points each) and for an overall score (with a maximum score of 50). The LEMS was defined as the sum of the motor function scores in the spinal segments lumbar level 2, lumbar level 3, lumbar level 4, lumbar level 5, and sacral level 1. A separate sum was obtained for the right and left sides (a maximum of 25 points each) and for an overall score (with a maximum score of 50).
Time Frame: Baseline to Day 3, Week 2, Week 4, Week 8, and Week 16 post dose.
Population: Total Motor Score (TMS) was assessed in the intent-to-treat (ITT) population, defined as all randomized participants who had at least 1 SCIM III evaluation and received at least 7 (partial or complete) IV bolus dose injections of the study drug in SUN13837 group or in Placebo group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Units on a scale
  Day 3 | 5.84 [1.56 to 10.12] | 1.20 [-2.95 to 5.35]
  Week 2 | 8.66 [3.55 to 13.77] | 4.04 [-0.89 to 8.97]
  Week 4 | 11.96 [6.19 to 17.72] | 6.35 [0.75 to 11.95]
  Week 8 | 14.81 [8.06 to 21.57] | 11.31 [4.69 to 17.93]
  Week 16 | 16.58 [9.40 to 23.76] | 14.07 [7.06 to 21.09]

4. Secondary Outcome: Self-Care and Mobility Subscale Scores of Spinal Cord Independence Measure, Version III (SCIM III) Score Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord Injury
Description: The SCIM III is a comprehensive rating scale that measures the ability of participants with spinal cord injury to perform everyday tasks. The SCIM III has 19 items that assess 3 domains, two of which are Self-care and Mobility. The self-care domain is a subscale of 6 items and scores range from 0 to 20 (higher scores indicate a better outcome). The mobility domain consists of 9 items with subscale scores range from 0 to 40 (higher scores indicate a better outcome). The score for the combined Self-Care and Mobility subscale ranges from 0 - 60 points; higher scores indicate a better outcome
Time Frame: Week 2, Week 4, Week 8, and Week 16 post dose.
Population: Self-Care and Mobility Subscale Scores were assessed in the intent-to-treat (ITT) population, defined as all randomized participants who had at least 1 SCIM III evaluation and received at least 7 (partial or complete) IV bolus dose injections of the study drug in SUN13837 group or in Placebo group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Score on a scale
  Week 2 | 5.76 [2.05 to 9.47] | 3.77 [0.18 to 7.35]
  Week 4 | 9.18 [4.81 to 13.56] | 6.45 [2.14 to 10.77]
  Week 8 | 14.70 [9.87 to 19.53] | 11.25 [6.47 to 16.03]
  Week 16 | 18.73 [13.43 to 24.03] | 15.02 [9.77 to 20.27]

5. Secondary Outcome: Upper Extremity Motor Scores (UEMS) of International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord
Description: The UEMS was defined as the sum of the motor function scores in the cervical spinal segments C5, C6, C7, C8, and T1. A separate sum was obtained for the right and left sides (a maximum of 25 points each) and an overall score of 0-50 with a maximum score of 50. A higher score indicates a better outcome.
Time Frame: Baseline to Day 3, Week 2, Week 4, Week 8, and Week 16 post dose.
Population: Upper Extremity Motor Scores (UEMS) were assessed in the intent-to-treat (ITT) population, defined as all randomized participants who had at least 1 SCIM III evaluation and received at least 7 (partial or complete) IV bolus dose injections of the study drug in SUN13837 group or in Placebo group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Units on a scale
  Day 3 | 2.08 [-0.14 to 4.31] | -1.24 [-3.45 to 0.98]
  Week 2 | 3.98 [1.50 to 6.46] | 0.59 [-1.83 to 3.02]
  Week 4 | 5.95 [3.40 to 8.50] | 1.73 [-0.79 to 4.24]
  Week 8 | 8.66 [5.94 to 11.38] | 3.83 [1.12 to 6.54]
  Week 16 | 9.92 [7.10 to 12.74] | 4.95 [2.17 to 7.73]

6. Secondary Outcome: Lower Extremity Motor Scores (LEMS) of International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord Injury
Description: The LEMS was defined as the sum of the motor function scores in the spinal segments lumbar level 2, lumbar level 3, lumbar level 4, lumbar level 5, and sacral level 1. A separate sum was obtained for the right and left sides (a maximum of 25 points each) and for an overall score with a maximum score of 50. A higher score indicates a better outcome.
Time Frame: Baseline to Day 3, Week 2, Week 4, Week 8, and Week 16 post dose.
Population: Lower Extremity Motor Scores (LEMS) were assessed in the intent-to-treat (ITT) population, defined as all randomized participants who had at least 1 SCIM III evaluation and received at least 7 (partial or complete) IV bolus dose injections of the study drug in SUN13837 group or in Placebo group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 27 | 28
Units on a scale
  Day 3 | 2.71 [0.15 to 5.28] | 3.22 [0.75 to 5.68]
  Week 2 | 3.66 [0.94 to 6.38] | 4.28 [1.67 to 6.88]
  Week 4 | 4.89 [1.82 to 7.96] | 5.36 [2.41 to 8.31]
  Week 8 | 5.08 [1.22 to 8.94] | 8.30 [4.53 to 12.08]
  Week 16 | 6.13 [1.80 to 10.46] | 9.96 [5.73 to 14.20]

7. Secondary Outcome: Incidence of Adverse Events Reported in ≥ 20% of Participants Following Treatment With SUN13837 Injection or Placebo in Adult With Acute Spinal Cord Injury
Description: The protocol defined an adverse event (AE) as any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Baseline up to approximately Day 182 post dose.
Population: The safety population was used to assess adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | SUN13837 | Placebo
Number analyzed (Participants) | 30 | 31
Participants
  Urinary tract infection | 21 | 23
  Pyrexia | 17 | 14
  Decubitus ulcer | 13 | 13
  Insomnia | 14 | 12
  Pneumonia | 9 | 17
  Nausea | 12 | 10
  Muscle spasticity | 12 | 9
  Neuralgia | 13 | 8
  Anxiety | 9 | 10
  Constipation | 7 | 11
  Leukocytosis | 8 | 10
  Depression | 8 | 9
  Musculoskeletal pain | 10 | 7
  Orthostatic hypotension | 9 | 8
  Anaemia | 5 | 11
  Respiratory failure | 8 | 7
  Muscle spasms | 8 | 6
  Headache | 9 | 4
  Rash | 9 | 4
  Blood creatine phosphokinase increased | 7 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to approximately Day 182 post dose.
Description: The protocol defined an adverse event (AE) as any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Serious AEs are summarized across the on-treatment and off-treatment periods by descending order in the SUN13837 group.
Arm/Group | SUN13837 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/30 | 2/31
Serious Adverse Events (participants affected / at risk) | 21/30 | 23/31
Other Adverse Events (participants affected / at risk) | 14/30 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUN13837 (N=30) | Placebo (N=31)
Anaemia (Blood and lymphatic system disorders) | 5 | 11
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1
Thyroiditis (Endocrine disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Euthanasia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 21 | 23
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 2 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 13 | 13
Withdrawal of life support (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 14 | 12
Pneumonia (Infections and infestations) | 9 | 17
Nausea (Gastrointestinal disorders) | 12 | 10
Muscle spasticity (Nervous system disorders) | 12 | 9
Neuralgia (Nervous system disorders) | 13 | 8
Anxiety (Psychiatric disorders) | 9 | 10
Constipation (Gastrointestinal disorders) | 7 | 11
Orthostatic hypotension (Vascular disorders) | 9 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 6
Headache (Nervous system disorders) | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUN13837 (N=30) | Placebo (N=31)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pyrexia (General disorders) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Neurogenic bladder (Nervous system disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Neurogenic bowel (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pseudomeningocele (Nervous system disorders) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Euthanasia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 3
Autonomic dysreflexia (Renal and urinary disorders) | 0 | 2
Alanin aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increase (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Spinal cord oedema (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Osteosynthesis (Skin and subcutaneous tissue disorders) | 0 | 1
Withdrawal of life support (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No